CLINICAL TRIAL: NCT00944047
Title: Abraxane and Trastuzumab Followed by Dose Dense Doxorubicin and Cyclophosphamide as Neoadjuvant Therapy in Invasive Breast Cancer With Low HER2 Expression (1+ or 2+ by IHC)
Brief Title: Evaluate Trastuzumab Plus Standard Chemotherapy Given Before Surgery in Breast Cancer Patients With Low HER 2 Expression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11368
Record Dates: First submitted 2009-07-16; First posted 2009-07-22 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: invasive breast cancer; HER2; primary breast cancer; neo-adjuvant therapy; Trastuzumab; Nab-paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Trastuzumab; Doxorubicin; Cyclophosphamide; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Arm (Experimental): Nab-paclitaxel, trastuzumab, doxorubicin, cyclophosphamide, Growth Factor Support, Surgery
  Interventions: Drug: nab-paclitaxel; Drug: trastuzumab; Drug: Doxorubicin; Drug: cyclophosphamide; Biological: Growth Factor Support; Procedure: Surgery

INTERVENTIONS:
Drug: nab-paclitaxel — 100 MG/M2 IV over 30 minutes once a week for 12 weeks
  Other Names: Abraxane
Drug: trastuzumab — 4 MG loading dose followed by 2 MG/KG every week for a total of 12 weeks
  Other Names: Herceptin
Drug: Doxorubicin — 60 MG/M2 every two weeks for a total of 4 cycles
  Other Names: Adriamycin
Drug: cyclophosphamide — 600 MG/M2 every 2 weeks for 4 cycles (administered with Doxorubicin above)
  Other Names: Cytoxan
Biological: Growth Factor Support — * All patients will receive pegfilgrastim 6.0 mg sc on Day #2 of each doxorubicin/cyclophosphamide neoadjuvant treatment cycle.
  * Erythropoetic growth factor support for fatigue/anemia will be allowed at the discretion of the treating physician.
Procedure: Surgery — * After completion of neoadjuvant therapy, patients will proceed with either modified radical mastectomy or lumpectomy.
  * All patients with pretreatment lymph node positive disease and positive sentinel lymph node will undergo complete axillary lymph node dissection.

SUMMARY:
The purpose of this study is to find out if there is a benefit of adding Herceptin (trastuzumab) to standard chemotherapy in this type of breast cancer.

DETAILED DESCRIPTION:
Neoadjuvant (primary) chemotherapy refers to chemotherapy given before surgery. Neoadjuvant chemotherapy has a number of potential advantages including increasing the chances for breast preservation at the time of surgery as well as it may improve the local control of the cancer. Several national breast cancer studies have shown that neoadjuvant chemotherapy was equal to chemotherapy given following surgery.

A standard treatment for stage II or Stage III invasive breast cancer with low HER2 expression is combination chemotherapyAdriamycin, Cytoxan,followed by a Taxane: given either before or after surgery), followed by surgery +/- radiation therapy.

The main purpose of chemotherapy however is to reduce the risk of recurrence of cancer and also make surgery more successful. HER2 is a receptor located on the surface of some cells. This receptor plays a role in regulating the growth of the cell, in addition to the growth of tumors. High levels of the HER2 receptor may predict those women who benefit from treatment with agents such as Herceptin that target HER2. Herceptin (Trastuzumab) is a drug that is effective both alone and in combination with standard chemotherapy. There is some data to suggest that patients whose tumors have low expression of the HER2 protein and are normal by FISH may also receive benefit from Herceptin.

ELIGIBILITY:
Inclusion Criteria:

* Female patient ≥ 18 years of age
* Histologically proven stage II or III adenocarcinoma of the breast
* Must be candidate for neoadjuvant treatment (Tumor size ≥ 2 cm, T2, T3, T4 and/or clinical N1 or N2).
* HER-2/neu 1+ or 2+ by immunohistochemistry
* Must have operable tumor.
* Performance status of 2 or better per SWOG criteria
* LVEF ≥ 55% by echocardiogram performed within 4 weeks prior to treatment initiation
* If patient of childbearing potential, pregnancy test is negative
* Patients with reproductive potential must use an effective method to avoid pregnancy for the duration of the trial.
* Adequate bone marrow function: ANC > 1500/mm3, platelet count > 100,000/mm3, and hemoglobin > 9 g/dL
* Adequate kidney function: serum creatinine of < 1.5mg/dl and/or creatinine clearance of > 60 mL/min
* Adequate hepatic function: transaminases < 2.5 x upper limit of normal and total bilirubin < 1.5 mg/dL
* Must be informed of the investigational nature of the study and must sign an informed consent in accordance with the institutional rules.
* Pretreatment lab values must be performed within 14 days of patient registration, and other baseline studies (with the exception of mammogram) must be performed within 30 days of patient registration.

EXCLUSION CRITERIA:

* Patient with metastatic breast cancer.
* Women with tumors that are HER-2 neu 0+ or 3+ by immunohistochemistry
* Women with HER 2 FISH amplified tumors (FISH ratio >2.2)
* Patients who have had prior endocrine therapy for > 4 weeks or chemotherapy for this breast cancer will be excluded.
* Locally advanced, inoperable tumors will be excluded.
* The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of drugs in this protocol or place the subject at undue risk for treatment complications.
* History of significant cardiac disease, cardiac risk factors or uncontrolled arrhythmias
* Ejection fraction < 55%
* Pregnancy or lactation
* Patients with inadequate laboratory values (as defined above) are excluded from study.
* Patients with NCI common toxicity criteria (CTC) grade 2 or greater peripheral neuropathy are excluded from study.
* Patients with active infection are excluded from study.
* Patients with concomitant or previous malignancies within the last 5 years, are excluded from the study. Exceptions include: adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, and ductal carcinoma in situ (DCIS).
* Patients with emotional limitations are excluded from study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-07; Primary Completion 2014-05 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qamar Khan, MD, Principal Investigator — University of Kansas Medical Center Cancer Center
Locations (2):
- United States (2):
  - Hays Medical Center, Hays, Kansas
  - University of Kansas Medical Center Cancer Center, Kansas City, Kansas

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: Nab-paclitaxel, trastuzumab, doxorubicin, cyclophosphamide, Growth Factor Support, Surgery
  nab-paclitaxel: 100 MG/M2 IV over 30 minutes once a week for 12 weeks
  trastuzumab: 4 MG loading dose followed by 2 MG/KG every week for a total of 12 weeks
  Doxorubicin: 60 MG/M2 every two weeks for a total of 4 cycles
  cyclophosphamide: 600 MG/M2 every 2 weeks for 4 cycles (administered with Doxorubicin above)
  Growth Factor Support: - All patients will receive pegfilgrastim 6.0 mg sc on Day #2 of each doxorubicin/cyclophosphamide neoadjuvant treatment cycle.
  - Erythropoetic growth factor support for fatigue/anemia will be allowed at the discretion of the treating physician.
  Surgery: -After completion of neoadjuvant therapy, patients will proceed with either modified radical mastectomy or lumpectomy.
  -All patients with pretreatment lymph node positive disease and positive sentinel lymph node will undergo complete axillary lymph node dissection.
Period: Overall Study
Arm/Group | Intervention Arm
Started | 32
Completed | 27
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Time Frame: 22 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 32
percentage of participants | 26

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | Intervention Arm
Serious Adverse Events (participants affected / at risk) | 5/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=32)
Febrile neutropenia (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Pain (General disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=32)
Allergic reaction (Immune system disorders) | 1 (1)
Rhinitis (Immune system disorders) | 3 (3)
Otitis, middle (Ear and labyrinth disorders) | 1 (1)
Blood - Other (Specify) (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5)
Leukocytes (Blood and lymphatic system disorders) | 2 (5)
Neutrophils (Blood and lymphatic system disorders) | 7 (10)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Vasovagal episode (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 27 (48)
Fever (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 16 (20)
Rigors/chills (General disorders) | 4 (4)
Weight gain (Investigations) | 4 (8)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 15 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 16 (28)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hot flashes (Endocrine disorders) | 5 (7)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 7 (11)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 16 (20)
Dehydration (Gastrointestinal disorders) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 15 (22)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 6 (6)
Esophageal mucositis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Heartburn (Gastrointestinal disorders) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 7 (9)
Nausea (Gastrointestinal disorders) | 25 (36)
Pharyngeal examination abnormal (Gastrointestinal disorders) | 1 (1)
Taste alteration (Gastrointestinal disorders) | 9 (11)
Tooth disorder (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (2)
Eye infection (Infections and infestations) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Infection - Other (Specify) (Infections and infestations) | 4 (7)
Infection, normal ANC, Lip/perioral (Infections and infestations) | 1 (1)
Infection, Urinary tract NOS (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 2 (3)
Otitis media (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 3 (5)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5)
Vaginal infection (Infections and infestations) | 2 (2)
Dermal change (Skin and subcutaneous tissue disorders) | 1 (1)
Edema limbs (General disorders) | 6 (8)
Edema: head and neck (General disorders) | 1 (1)
Creatinine increased (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 11 (12)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (7)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (6)
Depression (Psychiatric disorders) | 3 (3)
Dizziness (Nervous system disorders) | 7 (10)
Euphoria (Psychiatric disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 22 (27)
Tremor (Nervous system disorders) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (2)
Blurred vision (Eye disorders) | 1 (2)
Dry eye syndrome (Eye disorders) | 2 (2)
Watering eyes (Eye disorders) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 6 (7)
Anal pain (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest pain (Cardiac disorders) | 2 (2)
Chest wall pain (Cardiac disorders) | 2 (2)
Eye pain (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 10 (11)
Joint pain (Musculoskeletal and connective tissue disorders) | 8 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Pharyngolaryngeal pain (Gastrointestinal disorders) | 6 (7)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 4 (5)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Flu-like syndrome (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No